CLINICAL TRIAL: NCT01411774
Title: 1/2 D-cycloserine Augmentation of CBT for Pediatric OCD
Brief Title: D-cycloserine Augmentation of Cognitive Behavioral Therapy (CBT) for Pediatric Obsessive-compulsive Disorder (OCD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH093381 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-08-08 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-10

CONDITIONS: Obsessive-compulsive Disorder
Keywords: Obsessive-compulsive disorder; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Psychotherapy; Counseling; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive-behavioral therapy plus pill placebo (Active Comparator): This study arm involves the subject receiving 10 sessions of cognitive behavioral therapy with pill placebo taken 1 hour before the session.
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Pill placebo
- Cognitive-behavioral Therapy plus d-cycloserine (Experimental): This study arm involves the subject receiving 10 sessions of cognitive behavioral therapy with d-cycloserine taken 1 hour before the session.
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: d-cycloserine

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — All patients will receive 10 sessions of therapy over 8 weeks using the evidence-based CBT protocol in POTS (2004). Sessions 1-4 will be held twice weekly; sessions 5-10 will be held on a weekly basis. Sessions 1-3 do not include exposures and are devoted to psychoeducation, cognitive therapy, and hierarchy development. Sessions 4-10 involve E/RP exercises specific to each youth.
  Other Names: exposure and response prevention; psychotherapy; counseling
Drug: d-cycloserine — D-cycloserine will be encapsulated into 25mg with identical placebo capsules. Youth will take (1 or 2) DCS or identical placebo capsule 1 hour before sessions 4-10. A 0.7mg/kg dosage corresponds with dosages found to be effective in adult studies (50mg/estimated average adult weight of 70kg=.71mg/kg). Accordingly, doses for this study will be about 0.7mg/kg. Two dosing levels will be used based upon weight ranges to ensure comparable mg/kg levels: children weighing 25-45kg will be given a dosage of 25mg (~0.56-1.0 mg/kg/day), and children ≥46kg will be given 50mg provided in two 25mg capsules (~0.50-1.08mg/kg/day). Doses will be given 1 hour before therapy sessions 4-10.
  Arms: Cognitive-behavioral Therapy plus d-cycloserine
Drug: Pill placebo — The pill placebo will be identical to the active study medication in every respect (e.g., size, shape, number of capsules, etc.).
  Arms: Cognitive-behavioral therapy plus pill placebo

SUMMARY:
The investigators are conducting a randomized double-blind placebo-controlled study to assess the efficacy of d-cycloserine augmentation of cognitive-behavioral therapy for the treatment of pediatric obsessive compulsive disorder. This study represents an innovative approach in translating bench research findings into clinical research and testing a new approach for optimizing an effective psychotherapy with a safe non-psychotropic medication.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) affects 1-2% of children, runs a chronic course without treatment, and is associated with considerable functional impairment and poor quality of life. Although most patients with OCD respond to cognitive-behavioral therapy (CBT) or pharmacotherapy with a serotonin reuptake inhibitor (SRI), a substantial number of youth remain symptomatic after receiving these therapies. Pharmacological interventions with SRIs are only moderately efficacious, rarely produce remission, may be accompanied by side effects, and may not be an acceptable intervention to some parents. Medication augmentation strategies such as atypical antipsychotics are often used in children with partial response but have concerning metabolic effects and no systematic supporting efficacy or safety data. Although CBT is the gold standard treatment for pediatric OCD, not all patients benefit and the availability of skilled therapists is quite limited. Thus, there is a critical need for interventions to optimize treatment outcome in pediatric OCD. The primary mechanism in CBT is repeated and prolonged exposure to feared situations while abstaining from OCD rituals. This treatment is based on animal models of extinction of conditioned fears. Basic research on the neural circuitry underlying fear extinction led to the examination of d-cycloserine (DCS), a partial agonist at the NMDA receptor in the amygdala, as an agent capable of enhancing extinction learning. Following successful validation of this strategy in animals, six trials in adult humans - and one study in youth with OCD - provide support for DCS dosing as facilitating extinction learning that occurs during exposure-based psychotherapy. However, experts and agencies responsible for regulating drug indications in the US, including the FDA, recognize that safety and efficacy findings in adults should not be routinely extrapolated to children. The present study furthers pilot work on DCS to augment the effects of CBT in children with OCD. The investigators are conducting a double-blind randomized controlled trial, conducted at two sites, to examine the relative benefit of 10 psychotherapy sessions of which sessions 4-10 will be augmented with weight-adjusted doses of DCS (25/50mg) compared to CBT augmented with placebo. 150 youth (ages 7-17) with OCD will be randomly and evenly assigned to one of the two treatment conditions. The primary outcome will be change in OCD symptom severity assessed by independent evaluators. The study recruitment sites are the University of South Florida (USF) and Massachusetts General Hospital/Harvard Medical School (MGH). This study extends the first report of DCS augmentation in youth with anxiety disorder/OCD by conclusively investigating an innovative research approach that manipulates glutamatergic pathways to mediate improved outcomes of exposure-based psychotherapy based upon a translational model of the neurobiology of OCD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient youth with obsessive-compulsive disorder between the ages 7-17 years.
* A Children's Yale-Brown Obsessive-Compulsive Scale score ≥ 16
* Child has a Full Scale IQ≥85 as assessed on the WASI (within 90% CI).
* English speaking

Exclusion Criteria:

* Receiving concurrent psychotherapy or a past adequate trial of CBT for OCD. Families will have the option of discontinuing such services to enroll in the study.
* New Treatments: Initiation of an antidepressant within 12 weeks before study enrollment or an antipsychotic 6 weeks before study enrollment. No new alternative medications, nutritionals or therapeutic diets within 6 weeks of study enrollment.
* Established Treatment changes: Any change in established psychotropic medication (e.g., antidepressants, anxioloytics, stimulant, alpha agonist) within 8 weeks before study enrollment (6 weeks for antipsychotic). Alternative medications must be stable for 6 weeks prior to baseline.
* Current clinically significant suicidality or individuals who have engaged in suicidal behaviors within 6 months will be excluded.
* DSM-IV conduct disorder, autism, bipolar, schizophrenia or schizoaffective disorders; or substance abuse in past 6 months using all available information.
* Youth with hoarding symptoms that are their primary form of OCD.
* Weight less than 25.0 kg.
* Epilepsy, renal insufficiency, and current/past history of alcohol abuse.
* Pregnant or having unprotected sex [in females] as the effects of d-cycloserine on pregnancy are unknown.
* Presence of a significant and/or unstable medical illness that might lead to hospitalization during the study.
* Known d-cycloserine allergy.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - University of South Florida, St. Petersburg, Florida
  - Massachusetts General Hospital, Cambridge, Massachusetts

REFERENCES:
- [Background] Storch EA, Murphy TK, Goodman WK, Geffken GR, Lewin AB, Henin A, Micco JA, Sprich S, Wilhelm S, Bengtson M, Geller DA. A preliminary study of D-cycloserine augmentation of cognitive-behavioral therapy in pediatric obsessive-compulsive disorder. Biol Psychiatry. 2010 Dec 1;68(11):1073-6. doi: 10.1016/j.biopsych.2010.07.015. PMID 20817153

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive-behavioral Therapy Plus D-cycloserine: This study arm involves the subject receiving 10 sessions of cognitive behavioral therapy with d-cycloserine taken 1 hour before the session.
  Cognitive-behavioral therapy: All patients will receive 10 sessions of therapy over 8 weeks using the evidence-based CBT protocol in POTS (2004). Sessions 1-4 will be held twice weekly; sessions 5-10 will be held on a weekly basis. Sessions 1-3 do not include exposures and are devoted to psychoeducation, cognitive therapy, and hierarchy development. Sessions 4-10 involve E/RP exercises specific to each youth.
  d-cycloserine: D-cycloserine will be encapsulated into 25mg with identical placebo capsules. Youth will take (1 or 2) DCS or identical placebo capsule 1 hour before sessions 4-10. A 0.7mg/kg dosage corresponds with dosages found to be effective in adult studies (50mg/estimated average adult weight of 70kg=.71mg/kg).
Period: Overall Study
Arm/Group | Cognitive-behavioral Therapy Plus Pill Placebo | Cognitive-behavioral Therapy Plus D-cycloserine
Started | 72 | 70
Completed | 72 | 67
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-behavioral Therapy Plus Pill Placebo | Cognitive-behavioral Therapy Plus D-cycloserine | Total
Number analyzed (Participants) | 72 | 70 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72 | 70 | 142
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.54 (3.04) | 13.05 (2.93) | 12.93 (2.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 38 | 38 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 65 | 61 | 126
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 70 | 142

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive-Compulsive Scale.
Description: The Children's Yale-Brown Obsessive-Compulsive Scale measures the severity of OCD symptoms. There are 10 questions that are summed to arrive at a total score, with higher scores representing more severe OCD symptoms (scores range from 0-40).
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy Plus Pill Placebo | Cognitive-behavioral Therapy Plus D-cycloserine
Number analyzed (Participants) | 72 | 70
units on a scale | 13.53 [11.22 to 15.85] | 13.98 [11.6 to 16.36]

2. Secondary Outcome: Clinical Global Impression-Severity
Description: The Clinical Global Impression-Severity involves a trained clinician rating how severe the person's OCD symptoms are on a 0 to 6 scale, with higher scores corresponding to more severe symptoms. This rating only involves a clinician completing a single item.
Time Frame: 10 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cognitive-behavioral Therapy Plus Pill Placebo | Cognitive-behavioral Therapy Plus D-cycloserine
Number analyzed (Participants) | 72 | 70
units on a scale | 2.23 [1.89 to 2.56] | 2.28 [1.94 to 2.63]
Statistical Analysis 1: Comparison: Cognitive-behavioral Therapy Plus Pill Placebo vs Cognitive-behavioral Therapy Plus D-cycloserine; Test type: Superiority; p = .95, Mixed Models Analysis — p < .05 was the threshold of significance; Analysis for the outcomes used linear mixed-effects models, with treatment group as the between-participant factor and time as the within group factor

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Cognitive-behavioral Therapy Plus Pill Placebo | Cognitive-behavioral Therapy Plus D-cycloserine
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/70
Other Adverse Events (participants affected / at risk) | 0/72 | 0/70

LIMITATIONS AND CAVEATS:
We did not measure distress ratings within each exposure session, which prohibits examining whether D-cycloserine enhances outcomes when within-session distress reduction is achieved.

The sample was primarily of white race/ethnicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No